CLINICAL TRIAL: NCT05952908
Title: Effect of Quality Assured Simulation Training on Cardiac Device Implanter Skills
Brief Title: Effect of Simulation-based Procedure Training for Novice Cardiac Device Implanters Towards Implant Proficiency
Acronym: IMPROF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jorio Mascheroni (Other)
Responsible Party: Sponsor-Investigator, Jorio Mascheroni, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KUL0912559-001
Record Dates: First submitted 2023-06-30; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: Proficiency-based progression; Training; Simulation; Metrics
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proficiency-Based Progression training group (Experimental): Trainees in this group will follow the simulation-based implant training curriculum (same content/tools in both study arms) and they will be required to demonstrate a quantitatively defined proficiency benchmark at each training stage to be able to advance to the next stage (proficiency-based progression [PBP] approach).
  Interventions: Other: Proficiency-Based Progression simulation training
- Traditional training group (Active Comparator): Trainees in this group will follow the simulation-based implant training curriculum (same content/tools in both study arms) but they will not be required to demonstrate a quantitatively defined proficiency benchmark at each training stage to be able to advance to the next stage.
  Interventions: Other: Traditional simulation training

INTERVENTIONS:
Other: Proficiency-Based Progression simulation training — The simulation-based training curriculum is delivered - with proficiency requirements - with the aim of further enhancing trainees' implant skills, as an optional supplement to their academic/institutional training.
  Arms: Proficiency-Based Progression training group
Other: Traditional simulation training — The simulation-based training curriculum is delivered - without proficiency requirements - with the aim of further enhancing trainees' implant skills, as an optional supplement to their academic/institutional training.
  Arms: Traditional training group

SUMMARY:
This is an educational research study involving novice cardiac device implanters willing to further enhance their device implant skills through optional simulation-based training. The goal is to prospectively compare the effect of two different simulation-based training approaches on the quality of operators' implant performance in a simulated environment. The hypothesis is that a novel simulation training curriculum requiring trainees to demonstrate predefined proficiency benchmarks to advance (proficiency-based progression method) would generate superior performances compared to a traditional simulation training curriculum without proficiency requirements but identical content/tools. At the end of the instruction each trainee will perform a final simulated implant procedure which will be (anonymously) video-recorded and consequently scored by independent reviewers using previously validated intraoperative performance metrics. The effect of the two training approaches will be evaluated and performances compared by group for each metric independently.

DETAILED DESCRIPTION:
BACKGROUND: In cardiac device implant training, there is no common system to objectively assess trainees' ability to perform tasks at predetermined performance levels prior to in-vivo practice. Patients are potentially exposed to risks related to operators' early learning curve. A novel approach to enhance the learning outcome could be a metric-based, simulation training to proficiency. Such an approach to training is known as proficiency-based progression (PBP) and requires trainees to demonstrate a predefined proficiency benchmark, quantified by validated procedure performance metrics, before proceeding to the next stage of training. Published results in various domains of procedural medicine show that PBP trainees perform ~60% better compared to their non-PBP trained peers. This approach has never been tested for device implant training yet.

INTERVENTION: The training curriculum developed for the study purpose will cover a triple chamber device system implantation (i.e., cardiac resynchronization therapy = CRT) and will comprise two mandatory modules: a self-paced e-learning component and a peer-to-peer simulation-based component at a skill center. The content, the resources and the agenda of the training curriculum will be the same for both study groups; only the criteria for the trainees to proceed through the training stages will differ.

STUDY IMPLICATIONS: Compared to traditional simulation training, metrics-based training to proficiency may ensure a superior, consistent, objectively assessed target-level of operator's performance before they advance to (supervised) in-vivo practice.

ELIGIBILITY:
Inclusion Criteria:

* Physicians actively practicing cardiac device implantation at time of enrolment
* Minimum 20 pacemaker/defibrillator systems previously implanted as 1st operator
* Minimum 3 cardiac resynchronization therapy (CRT) systems previously implanted at least as 2nd operator
* Familiarity with English language (written and spoken)

Exclusion Criteria:

* Having previously implanted ≥ 200 CRT systems as 1st operator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Number of procedural Steps Completed in the final skills assessment (median per group) | 1 hour post-intervention
  Procedural Steps Completed is an intraoperative performance metric objectively assessed/scored from each trainee's (anonymous) simulated implant video-recording acquired at the end of the training as a final skills assessment. The analysis will compare the medians of each group.
Number of Errors in the final skills assessment (median per group) | 1 hour post-intervention
  Procedural Errors is an intraoperative performance metric objectively assessed/scored from each trainee's (anonymous) simulated implant video-recording acquired at the end of the training as a final skills assessment. The analysis will compare the medians of each group.
Number of Critical Errors in the final skills assessment (median per group) | 1 hour post-intervention
  Procedural Critical Errors is an intraoperative performance metric objectively assessed/scored from each trainee's (anonymous) simulated implant video-recording acquired at the end of the training as a final skills assessment. The analysis will compare the medians of each group.
Number of Errors All Combined (Errors + Critical Errors) in the final skills assessment (median per group) | 1 hour post-intervention
  Procedural Errors All Combined, represents the total amount of deviations from optimal performance (Errors + Critical Errors) and it's an overall indicator of performance quality. The analysis will compare the medians of each group.

SECONDARY OUTCOMES:
Procedure duration (min) in the final skills assessment (median per group) | 1 hour post-intervention
  Four procedural measures will be derived from video-recordings of the implant performances on the virtual reality simulator: Procedure duration, Fluoroscopy duration, Cineradiography duration, amount of Contrast Media injected. The analysis will compare the medians of each group (each variable is compared independently).
Fluoroscopy duration (min) in the final skills assessment (median per group) | 1 hour post-intervention
  Four procedural measures will be derived from video-recordings of the implant performances on the virtual reality simulator: Procedure duration, Fluoroscopy duration, Cineradiography duration, amount of Contrast Media injected. The analysis will compare the medians of each group (each variable is compared independently).
Cineradiography duration (s) in the final skills assessment (median per group) | 1 hour post-intervention
  Four procedural measures will be derived from video-recordings of the implant performances on the virtual reality simulator: Procedure duration, Fluoroscopy duration, Cineradiography duration, amount of Contrast Media injected. The analysis will compare the medians of each group (each variable is compared independently).
Contrast Media injected (ml) in the final skills assessment (median per group) | 1 hour post-intervention
  Four procedural measures will be derived from video-recordings of the implant performances on the virtual reality simulator: Procedure duration, Fluoroscopy duration, Cineradiography duration, amount of Contrast Media injected. The analysis will compare the medians of each group (each variable is compared independently).
Score obtained in the online knowledge test (percentage of correct answers per group, from 0 [minimum, worst outcome] to 100 [maximum, best outcome]) | 1 hour post-intervention
  At the completion of the online component of the training curriculum, trainees are required to take a summative knowledge test online. The scale title will be "Percentage of correct answers in the online assessment". The outcome will span from 0 [minimum, worst outcome] to 100 [maximum, best outcome].
Number of trainees per study group demonstrating the proficiency benchmark in the final assessment | 1 hour post-intervention
  The number of trainees per study group demonstrating the proficiency benchmark in the video-recorded performance at the end of the training curriculum.
Participants' satisfaction level at the end of the training curriculum (mean score per group on a Likert scale, from 0 [minimum, worst outcome] to 10 [maximum, best outcome]) | 3 hours post-intervention
  Participants' satisfaction level regarding the training received expressed on a Likert scale; feedback will be provided anonymously through the training evaluation forms filled at the end of the program. The scale title will be "Probability of recommending the curriculum to a peer". The outcome will span from 0 [minimum, worst outcome] to 10 [maximum, best outcome].

CONTACTS AND LOCATIONS:
Overall Officials: Jorio Mascheroni, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data that underlie results in publications, as well as data dictionaries, will be made available when access criteria are met.
Supporting Information: Study Protocol, SAP
Time Frame: Proposals may be submitted up to 36 months following article publication.
Access Criteria: Types of analyses: For individual participant data meta-analysis. Who can access the data: Investigators whose proposed used of the data has been approved by an independent review committee.

REFERENCES:
- [Derived] Mascheroni J, Stockburger M, Patwala A, Mont L, Rao A, Retzlaff H, Garweg C, Verbelen T, Gallagher AG. Effect of Metrics-Based Simulation Training to Proficiency on Procedure Quality and Errors Among Novice Cardiac Device Implanters: The IMPROF Randomized Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2322750. doi: 10.1001/jamanetworkopen.2023.22750. PMID 37651144